CLINICAL TRIAL: NCT05080218
Title: The SARS-CoV-2 Vaccine Response and Safety in Rheumatology Patients and the Influence of Temporary Interruptions in Immunomodulatory Therapy
Brief Title: COVID-19 VaccinE Response in Rheumatology Patients
Acronym: COVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jeffrey Curtis (Other)
Collaborators: University of Alabama at Birmingham (Other); University of Nebraska (Other); University of Pennsylvania (Other); AbbVie (Industry); Bristol-Myers Squibb (Industry); Novartis (Industry); Eli Lilly and Company (Industry); Pfizer (Industry); Illumination Health (Network)
Responsible Party: Sponsor-Investigator, Jeffrey Curtis, Physician Scientist, Foundation for Advancing Science Technology Education and Research
Organization: Foundation for Advancing Science Technology Education and Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COVER-Main
Record Dates: First submitted 2021-10-06; First posted 2021-10-15 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-06

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Spondylarthritis
Keywords: rheumatoid arthritis; COVID vaccine booster; spondyloarthritis; psoriatic arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylarthritis | interventions — upadacitinib; Abatacept; secukinumab; tofacitinib; Tumor Necrosis Factor Inhibitors; Etanercept; Certolizumab Pegol; Adalimumab; canakinumab; baricitinib; ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Treatment Interruption - UPA (Experimental): Treatment Interruption of Immunomodulatory Therapy for 2 Weeks at the time of COVID Vaccine Booster
  Interventions: Drug: Upadacitinib
- Treatment Continuation (No Intervention): Treatment Continuation of All Immunomodulatory Therapy at the time of COVID Vaccine Booster
- Treatment Interruption - ABA (Experimental): Treatment Interruption of Immunomodulatory Therapy for 2 Weeks at the time of COVID Vaccine Booster
  Interventions: Drug: Abatacept
- Treatment Interruption - TOF (Experimental): Treatment Interruption of Immunomodulatory Therapy for 2 Weeks at the time of COVID Vaccine Booster
  Interventions: Drug: Tofacitinib
- Treatment Interruption - SEC (Experimental): Treatment Interruption of Immunomodulatory Therapy for 2 Weeks at the time of COVID Vaccine Booster
  Interventions: Drug: Secukinumab
- Treatment Interruption - TNFi SQ (Experimental): Treatment Interruption of Immunomodulatory Therapy for 2 Weeks at the time of COVID Vaccine Booster
  Interventions: Drug: TNF Inhibitor
- Treatment Interruption - CAN (Experimental): Treatment Interruption of Immunomodulatory Therapy for 2 Weeks at the time of COVID Vaccine Booster
  Interventions: Drug: Canakinumab Injection
- Treatment Interruption - BAR (Experimental): Treatment Interruption of Immunomodulatory Therapy for 2 Weeks at the time of COVID Vaccine Booster
  Interventions: Drug: Baricitinib
- Treatment Interruption - IXE (Experimental): Treatment Interruption of Immunomodulatory Therapy for 2 Weeks at the time of COVID Vaccine Booster
  Interventions: Drug: Ixekizumab

INTERVENTIONS:
Drug: Upadacitinib — Hold UPA x 2 weeks at time of COVID booster
  Other Names: Rinvoq
  Arms: Treatment Interruption - UPA
Drug: Abatacept — Hold SQ ABA x 2 weeks at time of COVID booster
  Other Names: Orencia SQ
  Arms: Treatment Interruption - ABA
Drug: Secukinumab — Hold SEC x 2 weeks at time of COVID booster
  Other Names: Cosentyx
  Arms: Treatment Interruption - SEC
Drug: Tofacitinib — Hold TOF x 2 weeks at time of COVID booster
  Other Names: Xeljanz
  Arms: Treatment Interruption - TOF
Drug: TNF Inhibitor — Hold SQ TNFi x 2 weeks at time of COVID booster
  Other Names: Etanercept; Certolizumab; Golimumab SQ; Adalimumab
  Arms: Treatment Interruption - TNFi SQ
Drug: Canakinumab Injection — Hold CAN TNFi x 2 weeks at time of COVID booster
  Other Names: Ilaris
  Arms: Treatment Interruption - CAN
Drug: Baricitinib — Hold BAR x 2 weeks at time of COVID booster
  Other Names: Olumiant
  Arms: Treatment Interruption - BAR
Drug: Ixekizumab — Hold IXE x 2 weeks at time of COVID booster
  Other Names: Taltz
  Arms: Treatment Interruption - IXE

SUMMARY:
The COVID-19 VaccinE Response in Rheumatology patients (COVER) study is a multicenter randomized controlled trial designed to evaluate the efficacy and safety of a mRNA COVID-19 vaccine supplemental dose (booster) in patients with autoimmune conditions and to evaluate the impact of different immunomodulatory therapies on vaccine response. The investigators propose to recruit up to 1000- patients with autoimmune conditions who have a completed 2-dose regime of mRNA COVID-19 vaccine (>28 days prior) and who are planning to receive an additional dose of mRNA COVID-19 vaccine (i.e., booster). Participants in this study will be men and women 18 years and older with confirmed rheumatic disease, including psoriatic arthritis (PsA), axial spondyloarthritis (SpA) and rheumatoid arthritis (RA) who express a decision to receive the mRNA vaccination booster within 30 days post enrollment.

A primary objective of this study is to test the hypothesis that holding certain medications for a brief period of time around the time of COVID-19 vaccination might improve the response to the vaccine while not unduly having safety concerns with respect to the effects of their disease. During the study, participants using the immunomodulatory therapies described outlined in protocol will be randomized to temporarily hold (for 2 weeks) versus continue after they receive the COVID-19 vaccine supplemental dose. Patients who temporarily stop one of their medications for their autoimmune inflammatory disease may be at increased risk of flares of their autoimmune condition. If these occur, they are expected to occur within 2 - 4 weeks of treatment interruption. Detailed protocol outlines the hold schedules for the therapies to be randomized in this study.

DETAILED DESCRIPTION:
There is an urgent need to determine the immunogenicity and safety of COVID-19 vaccines in people living with rheumatic disease on immunomodulatory therapies. Given the experience with influenza, pneumococcal, shingles, and other vaccinations in rheumatic disease populations, it is clear that disease modifying therapies (DMARDs) and the immunomodulatory therapies used to treat immune-mediated inflammatory diseases have the capacity to blunt immune responses to vaccinations. A number of mostly small studies have examined the optimal management of DMARDs with regard to the timing of vaccination in order to maximize the immunogenicity of various vaccines, with immunogenicity serving as a lab-based proxy for clinical effectiveness. As various development programs near completion with regard to a vaccine for SARS-CoV-2 virus, it will be imperative to understand how best to vaccinate immunosuppressed patients, and in particular, to optimize vaccine response resulting from a supplemental (booster) dose in those patients using immunomodulatory biologic and targeted small molecule therapies. In concert with the American College of Rheumatology's (ACR) task force focused on developing COVID-19 vaccination guidance, the proposed real-world study will address major knowledge gaps that exist with the SARS-CoV-2 vaccination in rheumatic disease patients who have not been included in vaccine studies. Currently, the ACR task force for COVID-19 vaccination guidance recommends that patients temporarily (1-2 weeks) stop one of their medications for their autoimmune inflammatory disease. However, it is not known if stopping medications may increase risk of flares in their autoimmune condition. If these occur, they are expected to occur within 2-4 weeks of treatment interruption.

Approximately 1000 patients will be studied to address these questions about the vaccine response following supplemental (booster) dosing associated with the use of upadacitinib, baricitinib, abatacept, canakinumab, secukinumab, ixekizumab, tofacitinib, TNFi, guselkumab (conditional on resource availability), and ustekinumab (conditional on resource availability). Participants will be randomized to hold these treatments for two weeks, or to continue their medication without interruption.

Study Objectives and Hypotheses

To conduct a large, randomized controlled trial to evaluate SARS-CoV-2 vaccine supplemental dose response in a large population of patients with autoimmune conditions, designed to meet three specific objectives and aims:

1. Specific Aim 1: Evaluate the immunogenicity of SARS-CoV-2 vaccination in patients with autoimmune conditions, randomizing patients to briefly interrupt (i.e., hold for 2 weeks) versus continue various immunomodulatory therapies at the time that they receive a supplemental (i.e., booster) mRNA vaccine dose.

   * Primary outcome: quantitative measurement of immunoglobulin G (IgG) against SARS-CoV-2 using electrochemiluminescent (ECL) technology against the receptor binding domain (RBD) of spike protein.
   * Primary Hypothesis (H1a): The mean titer of anti-RBD IgG antibodies specific to SARS-CoV-2 measured post a third (booster) vaccine dose will be greater in patients randomized to temporarily hold (e.g., 2 weeks) versus those who continue immunomodulatory therapies.
   * Exploratory outcomes (with the randomized patients as the primary analysis population, and all patients as an additional analysis population):

     * Measures of cell-mediated immunity and neutralizing assay or other assays to be specified in the future (E1a).
     * Live-viral neutralization capacity post-vaccination (E1b).
     * Comparison of mean titer of anti-RBD IgG antibodies specific to SARS-CoV-2 measured post supplemental dose for each immunomodulatory therapy to be studied compared to tumor necrosis factor inhibitors.
     * Comparison of mean titer of anti-RBD IgG antibodies specific to SARS-CoV-2 measured post supplemental dose compared to general population.
     * Comparison of mean titer of anti-RBD IgG antibodies specific to SARS-CoV-2 measured post supplemental dose in patients receiving concomitant methotrexate (MTX) compared to patients not receiving concomitant MTX.
     * Comparison of mean titer of anti-RBD IgG antibodies specific to SARS-CoV-2 spike protein measured at baseline, by immunomodulatory medication received at the time of the initial vaccine series, and according to whether the immunomodulatory medication was held or not.
2. Specific Aim 2: Evaluate the safety and tolerability of SARS-CoV-2 vaccination in patients with different autoimmune conditions.

   * Secondary outcomes:

     * Flare and disease worsening of underlying autoimmune/inflammatory disease within 4 weeks of the supplemental vaccine dose.
     * Vaccine reactogenicity within 1 week of the supplemental vaccine dose.
     * Other safety events (e.g., allergic reactions, anaphylaxis, potential immune mediated adverse events).
   * Secondary Hypothesis #2 (H2b): the frequency of disease flare after the initial vaccine series and a supplemental vaccine dose will be higher in patients who hold immunomodulatory therapy compared to those who do not. Disease flare will be collected retrospectively through clinical measurements and patient reported outcomes for the initial vaccine series, and prospectively after receipt of the supplemental vaccine dose.
   * Exploratory outcomes: Comparison of circulating measures of inflammation (e.g., autoantibodies, cytokines, chemokines) between those holding and those continuing immunomodulatory therapy at the time of receipt of a supplemental dose of vaccine [conditional on funding availability].
3. Specific Aim 3 : Determine the clinical effectiveness of SARS-CoV-2 vaccination in patients with different autoimmune conditions and the subgroups of patients receiving different immunomodulatory therapies.

   * Exploratory outcome: clinical efficacy (i.e., clinically-recognized COVID infection events) as ascertained by active surveillance, as well as passive linkage to administrative health plan claims and electronic health record (EHR) data.

ELIGIBILITY:
Inclusion Criteria: *Patients must meet all of the inclusion criteria at the time of screening*

* Must have a rheumatology provider diagnosis of one or more of the following autoimmune inflammatory conditions:

  * Rheumatoid arthritis or adults previously diagnosed with Juvenile idiopathic arthritis (analyzed as a single category)
  * Psoriatic arthritis (PsA), Ankylosing spondylitis (ASp), or other Spondyloarthritis (SpA)
* Must have completed the 2-dose regimen of either of the two mRNA COVID-19 vaccines more than 28 days previous to enrollment
* Must be scheduled for an additional dose of mRNA COVID-19 vaccination booster (or with plans to schedule booster) within the next 30 days
* Must have a cell phone capable of receiving text messages, and/or a personal email address
* Currently receiving one of the medications described in Table 1
* Must be on stable immunomodulatory therapy for 8 weeks (with no dose changes, or interruptions > 2 weeks) prior to study enrollment. This would include both the qualifying immunomodulatory drug listed in Table 2, as well as any background immunomodulatory therapies (e.g. methotrexate, leflunomide) or glucocorticoids.
* Must be 18 years of age or older
* Must live in the United States.

Exclusion Criteria:

* • Already received a non-mRNA COVID-19 vaccine dose (J&J)

  * Any use in the past 90 days of a monoclonal antibody against COVID-19 (e.g., bamlanivimab, casirivimab, imdevimab)
  * Any known contraindication to COVID-19 vaccination, including allergic reaction to prior COVID-19 vaccination, and severe allergy to vaccine components (e.g., pegloticase)
  * Known HIV/AIDS or any other immunodeficient condition
  * Use of immunomodulatory therapy for any non-rheumatologic indication (e.g., organ transplantation)
  * Currently receiving radiation or chemotherapy for any type of malignancy.
  * Receipt of any immunization other than COVID-19 within two weeks prior to the COVID-19 vaccine supplemental dose
  * Significant underlying illness that would be expected to prevent completion of the study (e.g., life-threatening disease likely to limit survival to < 1 year)
  * Any other reason that, in the opinion of the site investigator, would interfere with required study related evaluations (e.g., uncontrolled disease flare, uncontrolled comorbidity)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 841 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Quantitative ratio post booster vs. pre-booster of IgG against SARS-CoV-2 using electrochemiluminescent (ECL) technology against the receptor binding domain (RBD) of spike protein, stratified by treatment arm | 6 weeks following COVID-19 vaccine booster
  Lab-based measure for immunogenicity (humoral immunity)

SECONDARY OUTCOMES:
Number of patients with score change beyond the minimal clinically important difference in the Rheumatoid Arthritis Flare Questionnaire (for patients with RA/PsA) and the BASDAI (Axial Spondyloarthritis), stratified by treatment arm | 6 weeks following COVID-19 vaccine booster
  Disease flare or worsening of underlying RA or SpA using a validated patient reported outcome
Number of patients with individual symptoms consistent with vaccine reactogenicity, as measured by the CDC Vsafe program, stratified by treatment arm | 6 weeks following COVID-19 vaccine booster
  Reactogenicity symptoms that confirm to the data collection methods by the Center for Disease Control as part of their VSafe program

OTHER OUTCOMES:
Number of patients with clinical COVID-19 infection, as initially self-reported by the patient, and confirmed by medical records, by treatment arm | 6 months following COVID-19 vaccine booster
  Relates to Specific Aim 3
Number of patients with clinical manifestations of new onset autoimmune disease and other pre-specified adverse events, as classified by CTCAE 4.0, by treatment arm | 6 months following COVID-19 vaccine booster
  e.g. Guillain Barre, pericarditis, myocarditis, relates to Specific Aim 2

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Curtis, MD MS MPH, Principal Investigator — Foundation for Advancing Science Technology Education and Research
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Illumination Health/Bendcare, Hoover, Alabama
  - Rheumatology Care Center, Hoover, Alabama
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Attune Health, Beverly Hills, California
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication, conditional on approval by the trial's steering committee
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the conclusion of the study.
Access Criteria: The investigators will share it with a secure FTP as requested by applicable parties.